CLINICAL TRIAL: NCT00002787
Title: Phase I Trial of Post Transplant Immunization With Autologous Myeloma Idiotype-KLH/GM-CSF In Myeloma Patients Following Autologous or Allogeneic Marrow or Stem Cell Transplantation
Brief Title: Vaccine Therapy in Treating Patients With Multiple Myeloma Who Have Undergone Stem Cell Transplantation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Maloney, David, Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Organization: Fred Hutchinson Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1104.00; NCI-2012-00669 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 1999-11-01; First posted 2004-05-21 (Estimated); Last update posted 2019-05-06 (Actual); Status verified 2019-05

CONDITIONS: Refractory Multiple Myeloma; Stage I Multiple Myeloma; Stage II Multiple Myeloma; Stage III Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — sargramostim; Granulocyte-Macrophage Colony-Stimulating Factor; aldesleukin; Interleukin-2

ARMS (1):
- Treatment (vaccine therapy) (Experimental): Patients receive autologous immunoglobulin idiotype-KLH conjugate vaccine combined with sargramostim SC in weeks 0, 2, 6, and 10 and sargramostim SC QD for three days following each vaccine injection. Some patients also receive aldesleukin SC daily from weeks 2-14.
  Interventions: Biological: autologous immunoglobulin idiotype-KLH conjugate vaccine; Biological: sargramostim; Biological: aldesleukin; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: autologous immunoglobulin idiotype-KLH conjugate vaccine — Given SC
  Other Names: autologous immunoglobulin idiotype-keyhole limpet hemocyanin conjugate vaccine; GTOP-99; Id-KLH; Id-KLH conjugate vaccine; recombinant Id-KLH
Biological: sargramostim — Given SC
  Other Names: GM-CSF; Leukine; Prokine
Biological: aldesleukin — Given SC
  Other Names: IL-2; Proleukin; recombinant human interleukin-2; recombinant interleukin-2
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
The purpose of this trial is to test the safety and immune response to four immunizations with this vaccine made from a protein produced by the patient's tumor. There is no guarantee or promise that this procedure will be successful

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety of multiple subcutaneous vaccinations with myeloma Id-KLH (idiotype-keyhole limpet hemocyanin) with GM-CSF (sargramostim) in post allogeneic transplant myeloma patients, or with GM-CSF +/- interleukin (IL)-2 (aldesleukin) in post autologous transplant myeloma patients.

II. To evaluate patients pre and post bone marrow transplantation (BMT) for evidence of endogenous idiotype specific immune response.

III. To characterize the time course, specificity and persistence of antibody and T cell immune response to myeloma idiotype and to KLH induced by myeloma Ig (Id) immunization.

IV. To clone, expand and characterize T cells specific for the tumor idiotype. V. Monitor myeloma involvement in bone marrow and serum paraprotein level following vaccination.

VI. Use stored patient samples to clone, expand, and characterize T cells specific for myeloma antigens other than idiotype and identify the antigens they recognize so that they can be used in future studies.

OUTLINE:

Patients receive autologous immunoglobulin idiotype-KLH conjugate vaccine combined with sargramostim subcutaneously (SC) in weeks 0, 2, 6, and 10 and sargramostim SC once daily (QD) for three days following each vaccine injection. Some patients also receive aldesleukin SC daily from weeks 2-14.

After completion of study treatment, patients are followed up every 3 months for 1 year and then every 6 months for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* ELIGIBILITY FOR VACCINE PREPARATION:
* Patients must have a diagnosis of multiple myeloma and be eligible for a Fred Hutchinson Cancer Research Center (FHCRC) treatment protocol using high dose therapy with syngeneic, allogeneic or autologous marrow or stem cell transplantation
* Pretransplant sera available with immunoglobulin A (IgA), immunoglobulin D (IgD), immunoglobulin E (IgE), immunoglobulin G (IgG), or immunoglobulin M (IgM) monoclonal paraprotein with a level of 1.5 grams/dl or greater identifiable on serum protein electrophoresis; eligibility for patients with pretransplant paraprotein levels of less than 1.5 gm/dl will be evaluated on an individual basis to determine whether purification of idiotype is feasible
* ELIGIBILITY FOR POST-TRANSPLANT IDIOTYPE VACCINATION:
* Successful isolation and production of an autologous idiotype vaccine from pre-BMT sera
* Greater than 60 days post BMT
* Achievement of a partial remission or greater (more than 75% reduction in serum paraprotein) for patients transplanted in relapse
* Stable absolute neutrophil count (ANC) > 1000
* Platelet count > 50,000 not requiring transfusions or growth factors
* Red blood cell (RBC) supportable to hematocrit (Hct) > 25 with less than 2 units of packed red blood cell (PRBC)/week
* Treatment with a stable dose of Interferon is allowed
* Karnofsky status > 60 percent
* Immunosuppression:

  * Off all corticosteroids
  * Either off all immunosuppressive medications or on a stable/tapering dose of cyclosporin or FK506 only

Exclusion Criteria:

* Graft-vs-host disease requiring treatment with corticosteroids
* Serum creatinine > 3.0
* Uncontrolled infection
* Disease progression
* Presence of medical complication that in the opinion of the investigators would result in inability to tolerate the vaccination protocol
* Patients with a history of serious adverse reactions to GM-CSF
* Patients with a history of serious adverse reactions to IL-2 will not receive concurrent IL-2 administration but may receive the Id-KLH vaccine with GM-CSF

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 1996-03; Primary Completion 2002-12 (Actual)

PRIMARY OUTCOMES:
Toxicities graded using the National Cancer Institute (NCI) Common Toxicity Criteria | Up to 2 years
  Descriptive statistics will be used to summarize changes from baseline in clinical laboratory parameters for each cohort.
Immune response | Up to 2 years
  Descriptive statistics will be used to summarize changes from baseline in clinical laboratory parameters for each cohort.

CONTACTS AND LOCATIONS:
Overall Officials: David Maloney, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (1):
- Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington, United States